CLINICAL TRIAL: NCT04360681
Title: Lofexidine Combined With Buprenorphine for Reducing Symptoms of Post-Traumatic Stress Disorder (PTSD) and Opioid Use Relapse in Veterans
Brief Title: Lofexidine Combined With Buprenorphine for Reducing Symptoms of PTSD and OU Relapse in Veterans
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); RTI International (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); USWM, LLC (dba US WorldMeds) (Industry); Foundation for Advancing Veterans' Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS170014-A6
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder; Opioid-use Disorder
Keywords: Opioid Use Disorder (OUD); Opioid; Opioid Use; Post Traumatic Stress Disorder (PTSD); Veteran
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Intervention Model Description: This is a Phase 2 randomized, double-blind, placebo-controlled, single-site, parallel groups, 12-week treatment study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To minimize bias, all participants will be screened for assurance that they meet study eligibility criteria. A placebo drug will be employed as the comparison group to active study drug and the study will be conducted in a double-blinded fashion in that both the participants and the site investigators and staff interacting with participants and assessing study outcomes will be blinded to treatment assignment. The only individuals at the site with assess to treatment assignment information will be the research pharmacists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lofexidine (LFX) (Experimental): LFX starting dosage is two 0.2 mg LFX tablet taken orally 2 times daily (i.e., 0.8 mg/day). At study visit 2 (Day 3), the dosage is increased to 1.2mg/day (3 tablets, BID). At visit 3 (Day 5), the dose is increased to the target dose of 1.6mg/day (4 tablets, BID). Participants enter the flexible dosing period at visit 4, at which point the LFX dose can be maintained at 1.6 mg/day or decreased to 1.2 mg/day based on symptoms and the clinical judgement of the investigator. The flexible dosing period extends through to visit 6, however, doses will be adjusted during the study as needed.
  Interventions: Drug: Lofexidine
- Placebo (PLB) (Placebo Comparator): A placebo drug will be employed as the comparison group to active study drug.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Lofexidine — BID dosing, and a max daily dose of 1.6 mg/day
  Other Names: LFX
  Arms: Lofexidine (LFX)
Drug: Placebo oral tablet — Placebo
  Other Names: PLB
  Arms: Placebo (PLB)

SUMMARY:
The overall objective of the proposed study is to determine if lofexidine (LFX) as an adjunct to buprenorphine (BUP) treatment improves symptoms of both opioid use disorder (OUD) and Post-Traumatic Stress Disorder (PTSD). Other study objectives are to compare the safety, tolerability, and efficacy of BUP treatment alone, to BUP treatment with adjunct LFX, on measures of OUD and PTSD symptoms in Veterans with both prognosis .

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the efficacy of Lucemyra™ (lofexidine; LFX), an alpha-2-adrenergic receptor (α2-AR) agonist, as a medication for the prevention of opiate relapse and the alleviation of post-traumatic stress disorder (PTSD) symptoms in opiate-dependent veterans.

Primary Endpoints :

For OUD:

Drug-Taking Behavior (% abstinent from illicit opioid use from Week 5 to Week 12 of the active treatment phase) is the primary efficacy endpoint for monitoring the effects of treatment on OUD, which is measured by both urine drug screen (UDS; opioids are detectable for 1-4 days) and timeline follow-back (TLFB) interviews of drug/alcohol use.

For PTSD:

The primary efficacy endpoint for monitoring the effects of treatment on PTSD symptoms is mean change scores on the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5), which is recommended by the Department of Veterans Affairs and the Department of Defense (VA/DoD) Clinical Practice Guideline as a quantitative measure of a patient's PTSD symptoms and response to treatment over time.

Secondary Endpoints:

For OUD:

Drug-Taking Behavior (≥ 80% abstinent between Week 5 to Week 12), treatment duration (days in treatment), and scores on the Subjective Opiate Withdrawal Scale (SOWS), the Clinical Opiate Withdrawal Scale (COWS), and the Opioid Craving Visual Analog Scale (OC-VAS) are secondary efficacy endpoints for monitoring the effects of treatment on symptoms on OUD.

For PTSD:

The secondary efficacy endpoints for monitoring the effects of treatment on core symptoms of PTSD are CAPS-5 change score (between screening and Week 12).

Population:

120 veteran participants will be recruited from within the MEDVAMC. The study population will consist of veterans diagnosed with OUD and potential or provisional PTSD who are seeking treatment.

Phase:

This is a Phase 2 randomized, double-blind, placebo-controlled, single-site, parallel groups, 12-week treatment study

Duration:

Enrollment period of 24 months. Participant duration is 18 weeks (consisting of 4 weeks screening, a 12-week treatment period, and a 2-week follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years of age, capable of reading and understanding English, and able to provide written informed consent (i.e. no persons who are imprisoned, of minor age, diagnosed with dementia, diagnosed with a terminal illness, or who otherwise require a surrogate to provide informed consent).
2. Be on a stable dose of BUP maintenance therapy for at least 7 days at the same maintenance dose. Veterans or non-Veterans who are not currently on a stable dose of BUP maintenance therapy will be referred to the Substance Dependence Treatment Program at the MEDVAMC or the Addiction Clinic at BTGH and invited to screen for this study once BUP treatment is stable.
3. Have a positive urine toxicology screen for BUP.
4. Has a previous diagnosis of PTSD documented in CPRS or meets criteria for current PTSD as assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).
5. Have hematology and chemistry laboratory tests within 3 months of study entry that are within normal (± 15%) limits, except liver function test results, which can be 5X the upper limit of normal.
6. Have a medical history and physical examination demonstrating no clinically significant contraindications for study participation within 3 months of study entry.

Exclusion Criteria:

1. DSM-5 criteria for substance use disorders (SUDs) other than OUD, nicotine, or cannabis, or stimulants [assessed by UDS and the Mini-International Neuropsychiatric Interview (MINI)].

   *Note that because the MINI assesses for SUDs over the past 12 months, potential participants will only be excluded if they both meet DSM-5 criteria for a SUD and have a positive UDS for that substance on study day 1. If a participant both meets DSM-5 criteria for a SUD and has a positive UDS at the screening visit, they will be informed that to be enrolled in the study they must have a negative UDS at their first study visit (i.e., prior to being enrolled).
2. Self-reported use of methadone in the last 14 days.
3. Be undergoing significant opioid withdrawal, as assessed by the COWS (defined as >12 on the COWS).
4. Increased risk of suicide that necessitates inpatient treatment or warrants therapy excluded by the protocol, and/or current suicidal plan, per investigator clinical judgement, based on interview and defined on the Columbia Suicidality Severity Rating Scale (C-SSRS).
5. Females of child-bearing potential must be using medically acceptable birth control (e.g. oral, implantable, injectable, or transdermal contraceptives; intrauterine device; double-barrier method) AND not be pregnant OR have plans for pregnancy or breastfeeding during the study.
6. Use of any of the following medications within 30 days prior to enrollment (self-report on Prior/Concomitant Medications (Meds) form):

   1. Benzodiazepines, barbiturates, or other CNS depressants
   2. Methadone or any other prescription analgesics, except BUP or BUP/naloxone
   3. Opioid antagonists such as naltrexone, except naloxone in combination with BUP
   4. Tricyclic antidepressants, which may reduce the efficacy of imidazoline derivatives
   5. Drugs that have been associated with QT prolongation, including:

   i. Antiarrhythmics: amiodarone, ajmaline, quinidine, disopyramide, procainamide, sotalol, ibutilide, dofetilide, etc.

ii. Antimicrobials

1. Fluoroquinolones: ciprofloxacin, levofloxacin, gatifloxacin, moxifloxacin, etc.
2. Macrolides: erythromycin, roxithromycin, azithromycin, clarithromycin, etc.
3. Antifungals: ketoconazole, itraconazole, etc. iii. Antipsychotics: haloperidol, thioridazine, ziprasidone, clozapine, quetiapine*, risperidone*, olanzapine, etc.

   f. Any other medications that might seriously and adversely interact with either LFX or BUP or have contraindication(s) to these medications
   * The following medications will be permissible at the discretion of the study physician:

<!-- -->

1. Bupropion a. Allowable dosage of up to 150mg daily (this is well below the therapeutic dose for depression, but is given for smoking cessation)
2. Quetiapine

   a. Allowable dosage 25mg -150 mg daily (typically given at night for sleep and well below the antipsychotic dosage of 400 mg or more)
3. Risperidone

   1. Allowable dosage 0.25mg- 1mg daily (below the antipsychotic dose of 2-8 mg daily) Prospective participants must be on a steady dose of the medication to be considered.

7. Prescription of any of the following medications within 30 days prior to enrollment (review of EDC patient chart):

a. Inducers or inhibitors of cytochrome P-450 3A4 (CYP3A4), the main metabolic enzyme of BUP: i. Antiretrovirals or other strong CYP3A4 inhibitors: boceprevir, cobicistat, conivaptan, danoprevir and ritonavir, elvitegravir and ritonavir, grapefruit juice, indinavir and ritonavir, itraconazole, ketoconazole, lopinavir and ritonavir, paritaprevir and ritonavir and ombitasvir and/or dasabuvir, posaconazole, ritonavir, saquinavir and ritonavir, telaprevir, tipranavir and ritonavir, troleandomycin, voriconazole, clarithromycin, diltiazem, idelalisib, nefazodone, nelfinavir, etc.

ii. Moderate CYP3A4 inhibitors: aprepitant, cimetidine, ciprofloxacin, clotrimazole, crizotinib, cyclosporine, dronedarone, erythromycin, fluconazole, fluvoxamine, imatinib, tofisopam, verapamil, etc.

iii. Anticonvulsants or other strong CYP3A4 inducers: carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's wort, etc.

8. Clinically significant abnormal ECG (such as second- or third-degree heart block, QTc interval ≥500 msec, uncontrolled arrhythmia), and/or history of a myocardial infarction.

9. Heart rate < 55 bpm or symptomatic bradycardia.

10. Systolic blood pressure < 90 mmHg, and/or diastolic blood pressure < 60 mmHg, and/or symptomatic hypotension.

11. Have a history of seizure disorder or severe traumatic brain injury (TBI); per the Ohio State TBI assessment.

12. Self-reported HIV/AIDS, active tuberculosis, and/or active syphilis.

13. Have significant hepatic, pancreatic (e.g., Type I diabetes), gastrointestinal or renal (that would affect absorption, metabolism or excretion of the study drug), endocrine, cardiac, neurological, psychiatric, pulmonary, hematologic, or other disorders (self-reported during Medical History assessment) that a study clinician believes would make study participation unsafe, treatment compliance difficult, or otherwise be determined by the PI to not be a good study candidate.

* The following conditions will be permissible at the discretion of the study physician:

  i. Type I &II diabetes- participants must meet the following criteria:

  1. Participants must be receiving MAT for at least 6 months 2. Hemoglobin A1c levels must be stable and relatively low 3 months prior to study entry and at the time of screening ii. Pancreatitis

  1. There must be 12 months between enrollment and last pancreatitis episode iii. Hepatitis

  1. Lab work submitted 3 months prior to study entry and at the time of screening should exhibit no elevations in liver functioning tests beyond 3X the upper limit of normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid Use | 12 weeks
  Drug-Taking Behavior (% abstinent from illicit opioid use from Week 5 to Week 12 of the active treatment phase) is the primary efficacy endpoint for monitoring the effects of treatment on OUD, which is measured by both urine drug screen (UDS; opioids are detectable for 1-4 days) and timeline follow-back (TLFB) interviews of drug/alcohol use.
PTSD Symptoms (Checklist) | 12 weeks
  The primary efficacy endpoint for monitoring the effects of treatment on PTSD symptoms is mean change scores on the PTSD Checklist for DSM-5 (PCL-5), which is recommended by the Department of Veterans Affairs and the Department of Defense (VA/DoD) Clinical Practice Guideline as a quantitative measure of a patient's PTSD symptoms and response to treatment over time.

SECONDARY OUTCOMES:
Opioid Withdrawal | 12 weeks
  Scores on opiate withdrawal scales, including the Subjective Opiate Withdrawal Scale (SOWS) and the Clinical Opiate Withdrawal Scale (COWS), are secondary efficacy endpoints. A lower total SOWS score (range: 0-64) indicates a more favorable clinical outcome. A COWS score of 5 to 12 is considered mild, 13 to 24 is moderate, 25 to 36 is moderately severe, and a score exceeding 36 is considered severe withdrawal. These scales are completed
PTSD Symptoms | 12 weeks
  CAPS-5 change score (between screening and Week 12) is a key secondary efficacy endpoint for PTSD

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D. Verrico, PhD, Principal Investigator — Baylor College of Medicine; Thomas R Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Congressionally Directed Medical Research Programs (CDMRP) has a policy to share and make available to the public the results and accomplishments of the activities that it funds. The Pharmacotherapies for Alcohol and Substance Abuse (PASA) Consortium plans to share de-identified data after final publication in a government-supported data repository